CLINICAL TRIAL: NCT06915662
Title: Pain Outcomes After Digital Amputation Using Tulavi Allay™ Nerve Cap: A Prospective Trial for Safety and Efficacy
Brief Title: Pain Outcomes After Digital Amputation Using Tulavi Allay™ Nerve Cap
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Tulavi Therapeutics,Inc. (Industry)
Responsible Party: Principal Investigator, Abhiram Bhashyam, Principal Investigator, Assistant Professor of Orthopaedic Surgery, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025P000828
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Neuroma; Neuropathic Pain
Keywords: Tulavi; Tulavi allay Nerve Cap; Neuroma; Neuropathic Pain; Digital Nerve Neuroma
MeSH Terms: conditions — Neuroma; Neuralgia

STUDY DESIGN:
Intervention Model Description: Surgeons will perform the procedure per their standard practice, but will use the allay™ Nerve Cap per the manufacturer's instructions to prevent potential symptomatic neuroma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Tulavi allay Nerve Cap (Experimental): Arm 1 will include patients who satisfy the inclusion criteria and consent to the study enrollment and procedure. Surgeons will perform the procedure per their standard practice, but will use the allay™ Nerve Cap per the manufacturer's instructions to prevent potential symptomatic neuroma.
  Inclusion Criteria:
  * Patients undergoing traumatic amputation of a single digit at MGB
  * English-speaking
  Exclusion Criteria:
  * Patients undergoing revision amputation or non-traumatic amputation
  * Patients under 22 years old
  * Patients who are pregnant and/or breastfeeding
  * Unable or unwilling to participate in a trial study
  All adult patients, satisfying the above inclusion and exclusion criteria, are eligible for enrollment in this study regardless of sex, race, or ethnicity. Vulnerable populations will not be recruited.
  Interventions: Device: Tulavi allay Nerve Cap

INTERVENTIONS:
Device: Tulavi allay Nerve Cap — The Tulavi allay Nerve Capfirst and only fully absorbable in situ forming technology designed to protect transected nerves, prevent axonal escape, and reduce the risk of neuroma formation.
  https://tulavi.com/allay-nerve-cap/

SUMMARY:
In 2016, one in five individuals in the United States (US) experienced chronic pain, and approximately 40% of them suffered from neuropathic pain. The physical and emotional burden on patients results in costs of billions of dollars annually. Digital amputations affect over 23,000 people each year in the US and may lead to neuropathic pain and neuroma formation in the transected nerves. Previous studies have reported a 6.6% incidence of symptomatic neuroma, and more than 60% of these patients require surgery to reduce the negative impact on their daily living activities.

To minimize neuroma formation after digital amputation, various techniques have been described, such as traction neurectomies (TN) and dorsal transpositions (DT), with and without nerve coaptation. However, it remains unclear whether these techniques improve patient-reported outcome measures in individuals undergoing this type of procedure. Previously published studies are descriptive in nature, focus on a single surgical technique, or include patients with established symptomatic neuromas. The only prospective trial on this topic was published in 2000 and compared two conventional techniques that have since been modified to better minimize neuroma formation or to reduce mechanical pressure by transposing the nerve ends to the dorsal aspect of the hand. However, that study used different scales to measure outcomes and did not incorporate aspects of pain that affect patients' emotional and social well-being.

Currently, two randomized controlled trials are enrolling patients. One compares surgical techniques for the treatment of neuroma rather than its prevention. The other excludes digits with injuries located distal to the interphalangeal joints. Both studies focus on more complex surgical techniques.

Given the extent of this problem, there has been recent innovation aimed at preventing neuroma formation. One promising product is the Tulavi Allay™ Nerve Cap, which has demonstrated encouraging results in basic science studies and anecdotally in early clinical use cases. In this study, the investigators have designed a prospective trial to assess the efficacy of the Tulavi Allay™ Nerve Cap when used to prevent symptomatic digital nerve neuroma following traumatic digital amputation.

DETAILED DESCRIPTION:
Background and Significance In 2016, one in five individuals in the United States (US) experienced chronic pain, and approximately 40% of them suffered from neuropathic pain. The physical and emotional burden on patients results in healthcare and societal costs of billions of dollars annually. Digital amputations affect over 23,000 people each year in the US and may lead to neuropathic pain and neuroma formation in the transected nerves. Previous studies have reported a 6.6% incidence of symptomatic neuroma, and more than 60% of these patients require surgery to reduce the negative impact on their daily activities.

To minimize neuroma formation after digital amputation, various techniques have been described, such as traction neurectomies (TN) and dorsal transpositions (DT), with and without nerve coaptation. However, it remains unclear whether these techniques improve patient-reported outcome measures in individuals undergoing this type of procedure. Previously published studies are largely descriptive, focus on a single surgical technique, or include patients with established symptomatic neuromas. The only prospective trial on this topic was published in 2000 and compared two conventional techniques that have since been modified to better minimize neuroma formation or reduce mechanical pressure by transposing nerve ends to the dorsal aspect of the hand. However, that study used heterogeneous outcome measures and did not assess the emotional and social impact of pain.

Currently, two randomized controlled trials (RCTs) are enrolling patients. One compares surgical techniques for the treatment of neuroma rather than its prevention. The other excludes patients with injuries to digits distal to the interphalangeal joint. Both studies focus on more complex surgical techniques.

Given the scope of this problem, there has been recent innovation aimed at preventing neuroma formation. One promising intervention is the Tulavi Allay™ Nerve Cap, which has demonstrated encouraging results in preclinical research and early clinical experience. In this study, the investigators have designed a prospective trial to assess the efficacy of the Tulavi Allay™ Nerve Cap in preventing symptomatic digital nerve neuroma following traumatic digital amputation.

General Description of Study Design This is a prospective trial. The investigators will enroll 20 patients. Questionnaires will be administered at the first post-operative appointment and again at 4-6 weeks, 3 months, 6 months, and 12 months post-operatively.

The following validated outcome measures will be used throughout patient participation:

Numerical Rating Scale (NRS): A standard 11-point pain scale (0 = no pain, 10 = worst possible pain). While no clinically significant change has been defined for digital amputation pain, studies on other chronic pain conditions have suggested that a reduction of 2 points represents a clinically meaningful difference.

Patient-Reported Outcomes Measurement Information System Pain Interference (PROMIS-PI): This instrument captures the impact of pain on emotional and social life. The investigators will use the PROMIS Pain Interference Computer-Adaptive Testing (PROMIS-PI CAT), which measures pain interference over the previous 7 days. PROMIS scores have a mean of 50 and a standard deviation (SD) of 10 in the reference population (US general population with pain).

Cold Intolerance Symptom Severity (CISS) Score: A six-item questionnaire (scored from 4-100), where each question ranges from 0 = no symptoms to 10 = most severe symptoms imaginable. The first question is not included in the final score. A score >50 is considered pathological cold intolerance.

Study Procedures

After surgery, patients who consent to participate will complete the following scales at five time points:

NRS pain score (0-10)

PROMIS-PI CAT (0-100)

CISS score (4-100)

These represent the primary quantitative outcomes and will be collected at:

First post-operative visit

1 month after surgery

3 months after surgery

6 months after surgery

12 months after surgery

Additional data will be collected at each visit using a custom questionnaire administered through REDCap (Research Electronic Data Capture):

Use of medication for neuropathic pain (Yes/No)

Engagement in desensitization physical therapy (Yes/No)

If patients are unable to attend an in-person visit or prefer remote follow-up, study staff will provide a REDCap survey link or administer the questionnaires by phone, depending on patient preference. Patients will have a two-week window to complete questionnaires. If questionnaires remain incomplete by the end of the two-week window, study staff will attempt contact for one additional week. After that, the data point will be marked as missing.

All enrolled patients will undergo surgery regardless of study participation. Remuneration is not applicable.

Study Termination Criteria:

Patient elects to withdraw from the study

Loss to follow-up (i.e., persistent missing data)

Regardless of study participation or withdrawal, patients will continue to receive standard clinical care. Physicians will remain accessible for consultation at all times.

Risks and Discomforts Surgical techniques for nerve stump management after digital amputation are currently selected based on surgeon preference, as there is no consensus on a superior method. All techniques aim to reduce the risk of symptomatic neuroma formation and related pain or discomfort.

The Tulavi Allay™ Nerve Cap has received De Novo classification by the U.S. Food and Drug Administration (FDA). Its use in this study does not expose patients to additional risk, as all patients already require nerve stump management as part of their surgical care.

While risks may vary depending on the cause of the amputation, potential implant-related risks include local tissue reaction or material failure. However, the hydrogel material used in the nerve cap is bioabsorbable. The product is provided as an in-kind research gift and will not result in additional cost to the patient.

Expected complications of both surgical techniques include: infection, injury to digital vessels, neuroma formation, hyperalgesia, cold intolerance, and neuropathic pain. No specific or unique complications related to the Tulavi Allay™ Nerve Cap have been reported.

A potential additional risk is the breach of confidentiality. To minimize this, all data will be collected electronically using REDCap, a secure, HIPAA (Health Insurance Portability and Accountability Act)-compliant, web-based platform hosted by Mass General Brigham (MGB) HealthCare Research Computing, through its Enterprise Research Infrastructure & Services (ERIS). Only study investigators and staff will have access to identifiable data. No paper-based records will be used. Once analysis is complete, all study data will be de-identified.

Benefits Currently, the most effective technique for preventing neuroma-particularly in terms of pain, cold intolerance, and pain interference-is not known. Therefore, there is no guaranteed individual benefit to participants. However, findings from this study may guide the development of future randomized controlled trials and improve neuroma management practices.

Statistical Analysis All statistical analyses will be conducted independently from Tulavi Therapeutics to avoid bias. The Principal Investigator (PI) has no financial conflict of interest.

A sample size of 20 patients has been established based on similar studies of other neuroma prevention techniques.

Data will be assessed for normality. Results will be reported as means and SDs for parametric data, medians and interquartile ranges for non-parametric data, and frequencies and percentages for categorical variables.

Relationships between explanatory variables and continuous outcomes will be assessed using simple linear regression and Pearson or Spearman correlation, as appropriate. For dichotomous explanatory variables, Mann-Whitney U or unpaired t-tests will be used. For categorical variables, Kruskal-Wallis and one-way ANOVA tests will be applied. In univariate analyses, statistical significance will be set at P ≤ 0.10.

Variables with statistically significant associations in univariate analysis will be included in a multivariable linear regression model to identify independent predictors of surgical outcomes, with significance set at P ≤ 0.05. If sample size limits the number of variables that can be included, the most clinically relevant and/or modifiable variables will be prioritized.

If imbalances between groups arise despite randomization, the investigators will consider stratification in the analysis. Based on existing literature and biological rationale, several variables may act as potential confounders or effect modifiers.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing traumatic amputation of a single digit at MGB
* English-speaking

Exclusion Criteria:

* Patients undergoing revision amputation or non-traumatic amputation Patients under 22 years old Patients who are pregnant and/or breastfeeding Unable or unwilling to participate in a trial study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Visual Analog / Numerical Rating Scale (VAS/NRS) Scores) | 12 months
  • Numerical Rating Scale (NRS): is a standard pain scale measured on a 11 point (0-10) where 0=no pain and 10=worst possible pain. There are no values defined as a clinically important difference for painful conditions in amputated digits, but previous studies on chronic painful conditions define a reduction of 2 points as a clinically important difference.
• Patient-Reported Outcomes Measurement Information System Pain Interference (PROMIS PI) | 12 months
  • Patient-Reported Outcomes Measurement Information System Pain Interference (PROMIS PI): this scale incorporates other aspects of pain that influence patient´s emotional and social life. We will use the most recent version PROMIS Pain Interference computer-adaptive testing (PROMIS IP CAT) that measures pain interference over the past 7 days. PROMIS scores have a mean of 50 and a SD of 10 in the reference population (U.S general population with a painful condition).
Cold Intolerance Symptom Severity score (CISS) | 12 months
  • Cold Intolerance Symptom Severity score (CISS) is a 6 questions scale with a possible total score from 4-100. Each question has a score of 0=no symptoms to 10=the most severe symptoms you can possibly imagine (the first question does not count for the final score). Previous studies suggested CISS>50 as a clinical cut-off for pathological cold intolerance.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Tulavi Therapeutics Inc. is providing the Tulavi allay™ Nerve Cap free of charge for this study. Data related to the safety and efficacy of the Nerve Cap, such as neuroma formation post-operatively, may be shared. Otherwise, no data will be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be available from the first enrolled patient (start date) until the final follow up of the last patient, 12 months after their procedure.
Access Criteria: The full-time research coordinator and principal investigator are responsible for adherence to all IRB policies and guidelines and for the accuracy and completeness of all forms, entries, and informed consent.
  Study data will be maintained in a locked filing cabinet and/or on password-protected computers. Questionnaires and self-reported responses will not become part of the subject's medical record. Hardcopies of study related data and forms will be stored in a lockable file cabinet. Only the investigators and study staff will have access to this information. Any magnetic or electronic information will be saved in password-protected computers to which only research coordinator and persons involved with the research project will have access. RED Cap, secure and HIPAA-compliant, will be used to collect questionnaire answers. All patient-identifiable information will be collected in a separate data log. The Principal Investigator oversees and monitors this process.

REFERENCES:
- [Background] Belcher HJ, Pandya AN. Centro-central union for the prevention of neuroma formation after finger amputation. J Hand Surg Br. 2000 Apr;25(2):154-9. doi: 10.1054/jhsb.2000.0372. PMID 11062573
- [Background] Reid DBC, Shah KN, Eltorai AEM, Got CC, Daniels AH. Epidemiology of Finger Amputations in the United States From 1997 to 2016. J Hand Surg Glob Online. 2019 Apr 1;1(2):45-51.
- [Background] Terwee CB, Peipert JD, Chapman R, Lai JS, Terluin B, Cella D, Griffiths P, Mokkink LB. Minimal important change (MIC): a conceptual clarification and systematic review of MIC estimates of PROMIS measures. Qual Life Res. 2021 Oct;30(10):2729-2754. doi: 10.1007/s11136-021-02925-y. Epub 2021 Jul 10. PMID 34247326
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Karcioglu O, Topacoglu H, Dikme O, Dikme O. A systematic review of the pain scales in adults: Which to use? Am J Emerg Med. 2018 Apr;36(4):707-714. doi: 10.1016/j.ajem.2018.01.008. Epub 2018 Jan 6. PMID 29321111
- [Background] Freniere BB, Wenzinger E, Lans J, Eberlin KR. Relocation Nerve Grafting: A Technique for Management of Symptomatic Digital Neuromas. J Hand Microsurg. 2019 Oct;11(Suppl 1):S50-S52. doi: 10.1055/s-0038-1677320. Epub 2019 Jan 4. PMID 31616128
- [Background] Taras JS, Tadley M, McCabe L. Dorsal Coaptation for the Treatment of Digital Neuroma. J Hand Surg Am. 2021 Jun;46(6):514.e1-514.e5. doi: 10.1016/j.jhsa.2020.10.027. Epub 2020 Dec 27. PMID 33375993
- [Background] Arnold DMJ, Wilkens SC, Coert JH, Chen NC, Ducic I, Eberlin KR. Diagnostic Criteria for Symptomatic Neuroma. Ann Plast Surg. 2019 Apr;82(4):420-427. doi: 10.1097/SAP.0000000000001796. PMID 30855369
- [Background] Lans J, Baker DJ, Castelein RM, Sood RF, Chen NC, Eberlin KR. Patient-Reported Outcomes following Surgical Treatment of Symptomatic Digital Neuromas. Plast Reconstr Surg. 2020 Mar;145(3):563e-573e. doi: 10.1097/PRS.0000000000006552. PMID 32097316
- [Background] Vlot MA, Wilkens SC, Chen NC, Eberlin KR. Symptomatic Neuroma Following Initial Amputation for Traumatic Digital Amputation. J Hand Surg Am. 2018 Jan;43(1):86.e1-86.e8. doi: 10.1016/j.jhsa.2017.08.021. Epub 2017 Sep 23. PMID 28951100
- [Background] Phillips CJ. The Cost and Burden of Chronic Pain. Rev Pain. 2009 Jun;3(1):2-5. doi: 10.1177/204946370900300102. PMID 26526940
- [Background] van Hecke O, Austin SK, Khan RA, Smith BH, Torrance N. Neuropathic pain in the general population: a systematic review of epidemiological studies. Pain. 2014 Apr;155(4):654-662. doi: 10.1016/j.pain.2013.11.013. Epub 2013 Nov 26. PMID 24291734
- [Background] Dahlhamer J, Lucas J, Zelaya C, Nahin R, Mackey S, DeBar L, Kerns R, Von Korff M, Porter L, Helmick C. Prevalence of Chronic Pain and High-Impact Chronic Pain Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Sep 14;67(36):1001-1006. doi: 10.15585/mmwr.mm6736a2. PMID 30212442
- [Background] Stjernbrandt A, Liljelind I, Nilsson T, Wahlstrom J. Defining abnormal cold sensitivity using the Cold Intolerance Symptom Severity questionnaire: a population study. J Hand Surg Eur Vol. 2021 Sep;46(7):731-737. doi: 10.1177/1753193421996221. Epub 2021 Mar 12. PMID 33709819
- See also: allay Nerve Cap webpage — https://tulavi.com/allay-nerve-cap/
- See also: Tulavi Therapeutics Inc. website — https://tulavi.com/